CLINICAL TRIAL: NCT07082192
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II/III Adaptive Clinical Study and Open-label Extension Study to Evaluate the Efficacy and Safety of Different Doses of CB03-154 in Adult Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study to Evaluate the Efficacy and Safety of Different Doses of CB03-154 in Adult Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Zhimeng Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB03-154-ALS201
Record Dates: First submitted 2025-07-11; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CB03-154 5mg (Experimental): Participants will receive CB03-154 5mg and Placebo 10mg orally once daily for 39 weeks.
  Interventions: Drug: Test drug CB03-154 5mg group
- CB03-154 10mg (Experimental): Participants will receive CB03-154 10mg and Placebo 5mg orally once daily for 39 weeks.
  Interventions: Drug: Test drug CB03-154 10mg group
- CB03-154 15mg (Experimental): Participants will receive CB03-154 15mg orally once daily for 39 weeks.
  Interventions: Drug: Test drug CB03-154 15mg group
- Placebo 15mg (Placebo Comparator): Participants will receive Placebo 15mg orally once daily for 39 weeks.
  Interventions: Drug: Placebo Group

INTERVENTIONS:
Drug: Test drug CB03-154 5mg group — One CB03-154 tablet (5mg/tablet) once daily.
  Arms: CB03-154 5mg
Drug: Test drug CB03-154 10mg group — Two CB03-154 tablets (5mg/tablet) once daily.
  Arms: CB03-154 10mg
Drug: Test drug CB03-154 15mg group — Three CB03-154 tablets (5mg/tablet) once daily.
  Arms: CB03-154 15mg
Drug: Placebo Group — Three Placebo tablets once daily.
  Arms: Placebo 15mg

SUMMARY:
The goal of this clinical trial is to learn if drug CB03-154 works to treat ALS in adults. It will also learn about the safety of drug CB03-154.

The main questions it aims to answer are:

* Does drug CB03-154 have an effect on delaying disease progression, improving function, and prolonging survival in adult ALS patients?
* What medical problems do patients have when taking drug CB03-154? Researchers will compare drug CB03-154 to a placebo (a look-alike substance that contains no drug) to see if drug CB03-154 works to treat ALS.

Participants (adult ALS patients) will:

* Take drug CB03-154 or a placebo every day for 39 weeks (an additional 39 weeks would be required if entering the open-label extension phase).
* Visit the clinic approximately every 2-3 months for checkups and tests, and there is also telephone follow-up in between.
* Keep a diary of daily medication (CB03-154 or other concomitant medications), and if there are any unplanned medications, the reason (disease or symptoms) also need be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the treatment plan and trial procedures of this study, and sign the written informed consent form.
2. Male or female, aged 18 to 65 years, inclusive.
3. The weight of subjects during the screening period must not be less than 45 kg, and the BMI must not be less than 18 kg/m2.
4. Diagnosed according to the Revised EI Escorial diagnostic criteria set by the World Federation of Neurology: definite ALS, probable ALS, lab supported probable ALS, or possible ALS.
5. Less than or equal to 24 months since ALS symptom onset at Screening, and estimated survival time of ≥1 year as per the Investigator's judgement.
6. Forced vital capacity (FVC) >80% of predicted value for gender, height, and age at Screening.
7. Able to swallow oral medication (tablets) at Screening as judged by the investigator.
8. For participants taking riluzole: Dose must be stable for at least 4 weeks prior to Screening and participant must be expected to remain on treatment for the duration of the trial. Participants receiving riluzole should maintain the same dose throughout the study.
9. Currently not receiving edaravone treatment or is in the schedule of edaravone treatment cycle. Participants receiving edaravone treatment must complete at least one cycle of treatment before the screening visit and continue stable dose edaravone treatment throughout the study.
10. Women of childbearing potential (WOCBP) must use an approved highly effective contraception for at least one menstrual cycle before the first dose of the investigational product and for at least 3 months after the last dose of the investigational product. Similarly, men must start using effective contraception before the first dose of the investigational product and continue for at least 3 months after the last dose of the investigational product, with no plans for procreation. Male participants cannot donate sperm for at least 3 months during the trial and after the last dose of the investigational product and female participants cannot donate or freeze eggs during the trial and for at least 3 months after the last dose of the investigational product.

Exclusion Criteria:

1. Significant cognitive impairment, mental disorders (such as schizophrenia, bipolar disorder), other neurodegenerative diseases (such as Parkinson's disease, Alzheimer's disease, frontotemporal dementia, etc.), substance abuse or other causes leading to neuromuscular weakness (such as myasthenia gravis), or other conditions that may interfere with the participants' participation in clinical study or, in the investigator's judgment, may interfere with outcome assessment or affect the completion of the trial.
2. Serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin>2.0× upper limit of normal at screening.
3. Estimated glomerular filtration rate <59 mL/min/1.73m2 at Screening (using the Cockcroft-Gault formula to calculate eGFR: eGFR (mL/min/1.73m2) = Ccr × 0.84 × 1.73 / BSA; Ccr (mL/min) = [(140 - age) × weight (kg)] / [72 × Scr (mg/dL)], females multiply the result by 0.85, and Scr is the serum creatinine; BSA (m2) = 0.007184 × weight (kg)^0.425 × height (cm)^0.725).
4. D-dimer>2.0× upper limit of normal or venous ultrasound of the lower limbs shows deep vein thrombosis at screening or a history of venous thrombosis.
5. Assistance with ventilation support or tracheostomy or tube feeding status or having a central venous catheter is required at screening.
6. A history of unexplained syncope, family history of syncope, or a history of convulsions or epilepsy (excluding the history of febrile seizures in childhood), or unstable medical condition, serious heart issues (e.g., corrected QTcF interval: males >450ms, females >470ms, torsades de pointes, NYHA class 3 or higher heart failure, myocardial infarction or unstable angina within 6 months prior to screening), lung, liver, kidney diseases, or tumors, or other clinically significant diseases or medical history (excluding ALS), participation in this study could threaten the safety of the participants.
7. Current clinically significant urinary retention, or current use of medications for urinary retention, or clinically significant abnormalities in residual urinary bladder ultrasound at screening.
8. Clinically significant ophthalmological abnormalities found in visual acuity examination (best corrected visual acuity), fundus photography, OCT examination, etc. during screening period, or clinically significant fundus lesions or retinopathy known or recorded in medical history.
9. Hepatitis B surface antigen (HBsAg) positive, or hepatitis C antibody (HCVAb) positive and hepatitis C virus ribonucleic acid (HCV-RNA) test higher than the lower limit of detection, or human immunodeficiency virus antibody (HIVAb) positive, or Treponema pallidum (TP) antibody positive (also judged as active infection by the investigator) at screening.
10. Severe infections (e.g., infectious pneumonia, sepsis) within 4 weeks prior to screening, or infections requiring hospitalization or intravenous administration of antibiotics, antiviral drugs, or antifungal medications, or chronic active bacterial infections (e.g., tuberculosis) deemed by the investigator to be unsuitable for participation in this trial.
11. Received Tofersen treatment before screening.
12. Significant risk of suicidality based on the Investigator's opinion or with an answer of "yes" on either item 4 or item 5 of the Suicidal Ideation Section of the Columbia Suicide Severity Rating Scale (C-SSRS) or any answer of "yes" within the Suicidal Behavior Section of the C SSRS within the 6 months before Screening.
13. Exposure to any other investigational medicinal product or product within 4 weeks or 5 half-lives of the investigational product (whichever is longer) prior to Screening; or exposure to monoclonal antibody drug within 6 months prior to Screening (or if the washout period at the time of screening has not reached more than 3 months), or had received cell therapy or gene therapy at any time in the past.
14. Treatment with CYP3A4 strong inducers or strong inhibitors prior to screening, and washout time of more than 5 half-lives of the drug was not reached before enrollment。
15. Pregnant, currently breastfeeding women or women with a positive pregnancy test at screening.
16. Known history of allergy to any component of the investigational medicinal product.
17. History of drug abuse within 12 months of Screening.
18. Anything else that, in the opinion of the Investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline to Week 39 in ALS Functional Rating Scale-Revised (ALSFRS-R).(Part A) Changes from Baseline to Week 78 in ALS Functional Rating Scale-Revised (ALSFRS-R).(Part B) | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)

SECONDARY OUTCOMES:
A joint rank analysis of function (Functional Rating Scale-Revised , ALSFRS-R) and survival(ALS/SURV)score at Week 39.(Part A) A joint rank analysis of function (Functional Rating Scale-Revised , ALSFRS-R) and survival(ALS/SURV)score at Week 78.(Part B) | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)
Change from Baseline and Slope of decline from Baseline in the Functional Rating Scale-Revised (ALSFRS-R) score at Weeks 8, 16, 28, 39, 51, 63 and 78. | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)
Change from Baseline and slope of decline in the Rasch Overall ALS Disability Scale (ROADS) score at Weeks 8, 16, 28, 39, 51, 63, and 78. | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)
Time from baseline to the earliest occurrence of 1 of the following events: first use of Permanent Assisted Ventilation (PAV) for >22 hours per day for >7 consecutive days OR death. | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)
Time from baseline to death. | From baseline to the entire period of double-blind period, assessed up to 39 weeks.
Change from Baseline in Forced Vital Capacity (FVC) at Weeks 8, 16, 28, 39, 51, 63 and 78. | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)
Change from Baseline in the Hamilton Depression Rating Scale, 17 item (HAMD-17) score at Weeks 8, 16, 28, 39, 51, 63, and 78. | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)
Change from Baseline in the Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) score at Weeks 8, 16, 28, 39, 51, 63 and 78. | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)
Change from Baseline on concentration of plasma Neurofilament Light Chain (NfL) at Weeks 8, 16, 28, 39, 51, 63 and 78. | From baseline to the entire period of double-blind period, assessed up to 39 weeks. (Part A) From baseline to the entire period of open-label extension, assessed up to 78 weeks. (Part B)